CLINICAL TRIAL: NCT06221098
Title: Study of Clinical Types and Treatment Outcomes of Pediatric Esotropia in Sohag University Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abeer Nasser Mazen, resident of ophthalmology department el helal hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-22-04-03
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Infantile Esotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- congenital esotropia (Active Comparator): will be defined as that type of esotropia with an onset prior to 6 months of age & characterized by a large stable angle
  Interventions: Procedure: bilateral medial rectus recession
- accommodative esotropia (Active Comparator): Fully accommodative esotropia will be defined as an esotropia which is controlled for distance and near with full hypermetropic correction. Partially accommodative esotropia will be defined as a reduction in the angle of esotropia of 10 dioptres or more for distance or near, using the full hypermetropic correctionAccommodative esotropia with convergence excess occurs when the near angle exceeded the distance angle by 15 dioptres or more when fixating an accommodative target, using the full hypermetropic correction.
  Interventions: Procedure: bilateral medial rectus recession
- non-accommodative esotropia (Active Comparator): neither congenital nor accommodative esotropia
  Interventions: Procedure: bilateral medial rectus recession

INTERVENTIONS:
Procedure: bilateral medial rectus recession — release muuscle from its original insertion and backword inserted in sclera
  Other Names: Monocular medial rectus (MR) recession and lateral rectus (LR) resection

SUMMARY:
Strabismus (or squint) is defined as the presence of misalignment between the visual axes of the 2 eyes presenting with deviation of the eyes. Strabismus is further subdivided into comitant (if the amount of misalignment between the 2 eyes remained equal in all directions of gaze) and incomitant (if the amount of misalignment varied in different directions of gaze). If the squinting eye was deviated inward, it is termed as a convergent squint or esotropia and if the squinting eye is deviated outward, it is termed as a divergent squint or exotropia. Pediatric esotropia may be congenital or acquired. Congenital esotropia is a well-defined entity with an onset prior to 6 months of age, characterised by a large stable angle, cross fixation, and a limited potential for binocular single vision. Acquired childhood esotropia may be paralytic or non-paralytic. The non-paralytic or concomitant type, which is neither congenital nor secondary to ocular pathology, can be divided into three main groups: (1) Accommodative esotropia, which may be fully accommodative, partially accommodative, or accommodative with convergence excess; (2) Non-accommodative esotropia; (3) Esotropia associated with neurological dysfunction, in particular cerebral palsy and hydrocephalus. The last group of esotropia will be excluded from our study. Pediatric strabismus must be treated early to maximize the potential for binocular vision and decrease the risk of amblyopia. Treatment goals include good vision in each eye (no amblyopia) and straight eyes (orthotropia). Both conditions are necessary to produce stereopsis, which is a third goal. Strabismus in children may result in undesirable appearance, amblyopia, impaired stereopsis, diplopia, and negative psychological effect.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children up to the age of 12 years.
2. Primary Concomitant convergent squint (1ry concomitant esotropia)
3. Candidate for surgical correction of squint

Exclusion Criteria:

* 1. Children with:

  1. Paralytic squint
  2. Consecutive esotropia
  3. Any neurological disorders e.g. hydrocephalus.
  4. History of previous squint surgery
  5. History of previous other ocular surgery (e.g. congenital cataract & glaucoma) 2. Children who missed follow up.

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
orthotropia | 6 months
  eye alignment
residual esotropia | 6months
  esotropia >10PD undercorrection
consecuative exotropia | 6 months
  exotropia > 10PD overcorrection

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohney BG. Common forms of childhood strabismus in an incidence cohort. Am J Ophthalmol. 2007 Sep;144(3):465-7. doi: 10.1016/j.ajo.2007.06.011. PMID 17765436
- [Background] Rubin SE, Nelson LB, Wagner RS, Simon JW, Catalano RA. Infantile exotropia in healthy children. Ophthalmic Surg. 1988 Nov;19(11):792-4. doi: 10.3928/0090-4481-19881101-07. PMID 3222041
- [Background] von Noorden GK. Bowman lecture. Current concepts of infantile esotropia. Eye (Lond). 1988;2 ( Pt 4):343-57. doi: 10.1038/eye.1988.65. PMID 3075563
- [Background] Mulvihill A, MacCann A, Flitcroft I, O'Keefe M. Outcome in refractive accommodative esotropia. Br J Ophthalmol. 2000 Jul;84(7):746-9. doi: 10.1136/bjo.84.7.746. PMID 10873987